CLINICAL TRIAL: NCT06213129
Title: Effect of Sodium and Ultrafiltration Profiling on Hemodynamic Stability, Interdialytic Weight Gain, and Intradialytic Complications.
Brief Title: Effect of Sodium and UF Profiling on Dialysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Neveen Hassan, MA Researcher, Assiut University
Other Study IDs: Na and UF profiling on ESRD
Record Dates: First submitted 2023-09-18; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Dialysis; Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Na and ultrafiltration profiling — Sodium and ultrafiltration profiling are method of dialysis in which dialysate sodium concentration and ultrafiltration rate are altered during the course of the dialysis session

SUMMARY:
The aim of this study is to evaluate the effects of sodium and UF profiling on hemodynamic stability, interdialytic weight gain, and intradialytic complications

DETAILED DESCRIPTION:
Sodium and ultrafiltration profiling are method of dialysis in which dialysate sodium concentration and ultrafiltration rate are altered during the course of the dialysis session.

Several sodium profiling methods are available. Increasing, decreasing, or alternating sodium concentrations may be used, although decreasing profiling has been the most accepted. The decrease in dialysate sodium concentration may be linear, stepwise, or exponential As different sodium profiling methods may have distinct impacts, different dialysis modalities may also affect the outcome of profiling. Although not as commonly used, hemodiafiltration HDF which utilizes convective clearance in addition to diffusion, may change the results of sodium profiling Such intervention alleviates the acute decline in intravascular volume during ultrafiltration UF as well as the decline in intradialytic plasma osmolarity and the consequent disequilibrium syndrome Sodium profiling enhances the internal plasma refill rate and helps to stabilize the blood pressure, thus decreasing the risk of Intra dialytic hypotension. It is imperative to limit or prevent intradialytic hypotension since it does not only affect the patient's comfort but also increases the risk of vascular access thrombosis, myocardial fibrosis and stunning, cardiovascular events, and mortality So it has potential benefits in terms of intradialytic morbidity and mortality as well as quality of life and long-term cardiovascular events; nevertheless, it may also predispose to interdialytic hypernatremia and increased interdialytic hypernatremia and interdialytic weight gain IDWG and hypertension. Fatigue and thirst have been reported with sodium profiling and the resulting sodium overload.

Another method to avoid intradialytic hemodynamic instability is UF profiling. In it, a larger portion of total UF volume is extracted during the first part of a dialysis session, after which the UF rate is decreased in order to maintain hemodynamic stability However, achieving a correct intradialytic sodium balance is a much more difficult task in clinical practice. With the advances in technology, automatic computer-based programs can be used today to calculate intradialytic sodium removal. These models use real-time data from patients and are being used to reach underdialysis sodium, weight in Kg, and blood volume targets. Such biofeedback systems enable to achieve sodium balance neutral sodium profile and UF profile automatically. Currently, there are various commercial dialysis systems that calculate dialysate and UF profiles with algorithms based on the prescribed decrease in body weight and sodium mass.

The aim of study to determine which specific profiling methods is more efficacious in preventing specific symptoms and which profiling method has the most utility in routine clinical practice. Furthermore, more qualitative data is warranted for subjective analysis of quality of life and personal well-being.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease patients.
* Patients on regular hemodialysis

Exclusion Criteria:

* Patients who refuse to contribute in this study.
* Hemodynamically unstable patients.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease on regular HD
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-08-28 (Estimated)

PRIMARY OUTCOMES:
systolic and diastolic blood pressure | 2 weeks
  The primary outcome is systolic blood pressure (80 _130)mmhg and diastolic blood pressure within range (60_80)mmhg, A blood pressure within this range is considered indicative of a better health outcome for the purposes of our research
Dialysis symptoms index | 2 weeks
  The Dialysis Symptom Index is a validated instrument to assess CKD-related unpleasant symptoms, and it is comprised of 30 questions about the presence of specifc symptoms For each question querying presence vs. absence of a specifc symptom, symptom severity is assessed using a five-point Likert scale, with each response ranging from 0 to 4 (i.e., a response of "0" indicates "no," whereas a response of "4" indicates "yes: very much"). The minimum-maxi- mum Dialysis Symptom Index score ranges from 0 to 120,with higher scores indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: youssef Saleh, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coli L, La Manna G, Dalmastri V, De Pascalis A, Pace G, Santese G, Stefanio C, Ursino M, Zaca F, Stefoni S. Evidence of profiled hemodialysis efficacy in the treatment of intradialytic hypotension. Int J Artif Organs. 1998 Jul;21(7):398-402. PMID 9745994